CLINICAL TRIAL: NCT02731573
Title: A Phase Ib/II Prospective, Multicenter, Two Part Study; Part 1 - Open Label, Single Arm & Part 2 Randomized, Single-blinded (Study to Assess Safety and Efficacy of D-PLEX Concomitantly With Standard of Care vs. Standard of Care Alone in the Prevention of Primary Sternal Infection Post Cardiac Surgery.
Brief Title: Safety and Efficacy of D-PLEX in the Prevention of Sternal Infection Post Cardiac Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PolyPid Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: D-PLEX -301 study
Record Dates: First submitted 2016-03-24; First posted 2016-04-07 (Estimated); Last update posted 2019-01-22 (Actual); Status verified 2018-06

CONDITIONS: Postoperative Wound Infection Superficial Incisional; Postoperative Wound Infection Deep Incisional Surgical Site
Keywords: Mediastenitis

STUDY DESIGN:
Intervention Model Description: Phase Ib/II, Prospective, Multicenter, Two part study; Part 1 Open Label, Single arm & Part 2 Randomized, Single-blinded, D-PLEX Concomitantly with Standard Of Care vs. Standard of Care alone.
  Study population include subjects above the age of 18 years, that undergoing cardiac surgery through mid-sternotomy, including patients with high risk of infection, such as diabetes (Insulin and/or non-insulin dependent), patients with Peripheral Vascular Disease (PVD), Chronic Obstructive Pulmonary Disease (COPD), heavy smokers, Bilateral Mammary artery harvesting, and subjects administered chronic steroid treatment.
  Subjects who meet the eligibility criteria and provide signed informed consent, will be enrolled into the study and will be treated with D-PLEX concomitantly with standard of care (part 1) or randomized 2:1 to D-PLEX concomitantly with standard of care vs. standard of care only (part 2).
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment arm (Experimental): Subjects who meet the eligibility criteria and provide signed informed consent, will undergo open heart surgery according to standard of care with treatment by D-PLEX.
  Interventions: Drug: D-PLEX; Procedure: Open heart surgery
- Control arm (Other): Subjects who meet the eligibility criteria and provide signed informed consent, will undergo open heart surgery according to standard of care.
  Interventions: Procedure: Open heart surgery

INTERVENTIONS:
Drug: D-PLEX — D-PLEX will be administered as a single application during the open heart surgery (index procedure) immediately prior to sternal closure, as an adjunct to the standard care.
  Arms: Treatment arm
Procedure: Open heart surgery — Subject will undergo open heart surgery according to standard of care
  Other Names: SOC

SUMMARY:
This study is aimed to assess the anti-infective efficacy of D-PLEX over a period of 3 months post operation as well as the safety over a period of 6 months, by preventing sternal infection post cardiac surgery in patients above the age of 18, including high risk patients for infection. This study is a 2 parts study: part 1 is a single arm, part 2 is randomized controlled study.

DETAILED DESCRIPTION:
D-PLEX is a new formulation of extended controlled release Doxycycline.

Subjects who meet the eligibility criteria and provide signed informed consent, will be enrolled into the study and will be treated with D-PLEX concomitantly with standard of care.

D-PLEX will be administered as a single application during a cardiac surgery (index procedure) immediately prior to sternal closure, as an adjunct to the standard care.

The study will assess the efficacy and safety of the controlled release antibiotic (doxycycline) by the reduction in the number of sternal infections observed during the treatment period in any subject above the age of 18 years, including patients with high risk for infection.

Additional follow up for prolonged safety assessments only, will be done as follows until 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female above 18 years old
2. Female of childbearing potential should have a negative serum pregnancy test prior to index procedure.

   Note: All female of childbearing potential must agree to use a highly effective method of contraception (such as double barrier, oral or parenteral hormonal, intrauterine device and spermicide) consistently and correctly for the duration of the study.
3. Subjects undergoing elective or urgent cardiac surgery, who are preoperative stable hemodynamically.
4. Subjects with (20≤BMI≤40)
5. Subjects who sign a written informed consent.

Exclusion Criteria:

1. Received any investigational drug within 30 days of start of study or within 5½ half-lives (pharmacokinetic or pharmacodynamics) prior to enrollment (whichever is longer).
2. Are ineligible to receive treatment with:

   * Any preoperative active significant infection
   * Antibiotic sensitivity to Doxycycline and/or tetracycline family of drugs
   * Known allergies to more than 3 substances.(Patients should fill the allergy questioners during the enrolment process)
   * History of allergic/hypersensitivity reaction to any substance having required hospitalization and/or treatment with intra-venous steroids/epinephrine or in the opinion of the investigator the patient is at high risk of developing severe allergic / hypersensitivity reactions.
   * History of uncontrolled Asthma (GINA III-IV)
   * History of chronic urticaria
3. Pregnant or breastfeeding women.
4. Subjects who have taken oral or IV doxycycline during the last 4 weeks prior to screening.
5. Subjects who undergo cardiac/open chest surgeries, which are classified as emergency.
6. Immunocompromised subjects from any reason, at screening.
7. Subjects that undergone TIA/ CVA within the last 3 months prior to enrollment.
8. Subjects that previously underwent any cardiac surgery through mid-sternum.
9. In the opinion of investigator, subject is not eligible to participate in the study due to a cognitive status, medical condition or medication status (other than items listed above)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Sternal Infection identified within 90 days post-cardiac surgery. Primary sternal infection as measured by the proportion of subjects with at least 1 identified primary sternal infection within 90 days post-cardiac surgery. | Within 90 days post-cardiac surgery.
  Decrease of infection rate as measured by the proportion of subjects with at least 1 identified sternal infection within 90 days post-cardiac surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Erez Kachel, MD, Principal Investigator — Sheba MC
Locations (5):
- Israel (5):
  - Soroka Medical Center, Beersheba
  - Rambam Medical Center, Haifa
  - Assuta Medical Center, Tel Aviv
  - Sheba Medical Center, Tel Litwinsky
  - Poriya Medical Center, Tiberias

IPD SHARING:
Plan to Share IPD: No